CLINICAL TRIAL: NCT06476899
Title: A Practical Clinical Study Comparing the Fixed-cycle Regimen Containing Orelabrutinib With BTKi Monotherapy in Previously Untreated CLL/SLL
Brief Title: A Practical Clinical Study Comparing the Fixed-cycle Regimen Containing Orelabrutinib With BTKi Monotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fei Li (Other)
Responsible Party: Sponsor-Investigator, Fei Li, Chief physician, The First Affiliated Hospital of Nanchang University
Organization: The First Affiliated Hospital of Nanchang University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PragmatiCLL
Record Dates: First submitted 2024-06-19; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: CLL/SLL
MeSH Terms: interventions — orelabrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed regimen (Experimental): orelabrutinib + FCR/BR
  Interventions: Drug: orelabrutinib; Drug: FCR/BR
- Control (Active Comparator): BTKi chosen by doctors
  Interventions: Drug: BTK inhibitor

INTERVENTIONS:
Drug: orelabrutinib — orelabrutinib tablets
  Arms: Fixed regimen
Drug: FCR/BR — FCR/BR
  Arms: Fixed regimen
Drug: BTK inhibitor — BTK inhibitor choose by physican
  Arms: Control

SUMMARY:
Prospective, interventional, and practical clinical studies

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years, with no gender restrictions;
* Patients with CLL/SLL who meet the iwCLL2018 diagnostic criteria;
* Indications for treatment
* ECOG performance score of 0-2;
* Patients are untreated or have not received standardized treatment
* Before the trial screening, the subject or their legal representative voluntarily signs a written informed consent form, indicating that they understand the purpose of the study and the necessary research steps, and are able to comply with the protocol and follow-up.

Exclusion Criteria:

* Has been diagnosed or treated for malignancies other than CLL (including active central nervous system lymphoma) within the past year;
* there is clinical evidence of Richter transformation;
* Participant cannot receive or plan to receive another treatment during study participation
* Other conditions that the investigator considers inappropriate for participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-24 (Estimated); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
TTNTD rate at 30 months | 30 months
  The proportion of time from the start of treatment to the start of the next treatment or death over a period of 30 months

SECONDARY OUTCOMES:
PFS | 3 years
  The time from the start of treatment to the point when the disease progression or death is confirmed by the investigator

IPD SHARING:
Plan to Share IPD: No